CLINICAL TRIAL: NCT02293837
Title: Preserving Beta-Cell Function With Tocilizumab in New-onset Type 1 Diabetes (ITN058AI)
Brief Title: Tocilizumab (TCZ) in New-onset Type 1 Diabetes
Acronym: EXTEND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); PPD Development, LP (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT ITN058AI
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes Mellitus; New-onset Type 1 Diabetes Mellitus; T1DM; T1D
Keywords: interleukin-6 (IL-6) receptor inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — tocilizumab; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tocilizumab (TCZ) + SOC (Experimental): Subjects will receive intravenous (IV) infusions of either 8.0 mg/kg (body weight ≥30 kg) or 10.0 mg/kg (body weight <30kg) tocilizumab every 4 weeks for 24 weeks. Participants will also receive standard intensive diabetes management (in accordance with the American Diabetes Association guidelines [Standard of Care, SOC])
  Interventions: Drug: Tocilizumab (TCZ); Other: Standard of Care
- Tocilizumab Placebo Group + SOC (Placebo Comparator): Subjects will receive IV infusions of either 8.0 mg/kg (body weight ≥ 30kg) or 10.0 mg/kg (body weight <30kg) placebo every 4 weeks for 24 weeks. Participants will also receive standard intensive diabetes management (in accordance with the American Diabetes Association guidelines [Standard of Care, SOC])
  Interventions: Drug: Placebo; Other: Standard of Care

INTERVENTIONS:
Drug: Tocilizumab (TCZ) — Subjects assigned to this group will receive tocilizumab intravenous (IV) infusions of either 8.0 mg/kg (body weight ≥ 30kg) or 10.0 mg/kg (body weight <30kg) every 4 weeks for 24 weeks.
  Other Names: Actemra®
  Arms: Tocilizumab (TCZ) + SOC
Drug: Placebo — Subjects assigned to this group will receive placebo intravenous (IV) infusions of either 8.0 mg/kg (body weight ≥ 30kg) or 10.0 mg/kg (body weight <30kg) every 4 weeks for 24 weeks.
  Other Names: Placebo for Tocilizumab
  Arms: Tocilizumab Placebo Group + SOC
Other: Standard of Care — Participants will also receive standard intensive diabetes management (in accordance with the American Diabetes Association guidelines [Standard of Care, SOC])
  Other Names: SOC

SUMMARY:
Type 1 diabetes mellitus (T1DM) is an autoimmune disease. Based on previous research, study doctors think that giving medicines to affect the immune system soon after diabetes is diagnosed may stop, delay or decrease the destruction of beta cells, resulting in better glucose control.

Researchers believe that tocilizumab could have some effect on the cells in the immune system that are thought to be involved in the development of type 1 diabetes. This study will test whether tocilizumab can help preserve or delay destruction of remaining beta cells in people recently diagnosed type 1 diabetes.

DETAILED DESCRIPTION:
Staggered enrollment is planned for this trial.

Prior to initiating the study in the pediatric age group (6-17 years old), 30-99 eligible adults (ages 18-45 years) will be randomized 2:1 to tocilizumab or placebo, respectively. Once the first thirty adult participants have completed 12 weeks of treatment, the FDA and Data and Safety Monitoring Board (DSMB) will review available data (e.g., interim analysis) to weigh potential risks and benefits before opening the trial to pediatric participants.

As of ≥ May 15, 2017: Study enrollment limited to participants ages 6 to 17 years inclusive.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 6-45 years*

   -*Current Institutional Review Board (IRB)-approved age eligibility criteria is restricted to subjects 6 to 17 years of age at time of study enrollment
2. Diagnosis of type 1 diabetes mellitus (T1DM), using the American Diabetes Association T1DM criteria, within 100 days of study enrollment
3. Positive for at least one diabetes-related autoantibody, including but not limited to:

   1. Glutamate decarboxylase (GAD-65)
   2. Insulin, if obtained within 10 days of the onset of exogenous insulin therapy
   3. Insulinoma antigen-2 (IA-2)
   4. Zinc transporter-8 (ZnT8)
4. Peak stimulated C-peptide level ≥ 0.2 pmol/mL following a mixed-meal tolerance test (MMTT) conducted at least 21 days from diagnosis and within 37 days of randomization (V0)
5. Signed informed consent (and informed assent of minor, if applicable).

Exclusion Criteria:

1. Severe reaction or anaphylaxis to human, humanized or murine monoclonal antibodies
2. History of malignancy or serious uncontrolled cardiovascular, nervous system, pulmonary, renal, or gastrointestinal disease, or significant dyslipidemia
3. Any history of recent serious bacterial, viral, fungal, or other opportunistic infections
4. Have serologic evidence of current or past HIV (Human immunodeficiency virus), Hepatitis B, or Hepatitis C
5. Positive QuantiFERON Tuberculosis (TB) test, history of TB, or active TB infection
6. Active infection with Epstein-Barr virus (EBV) as defined by EBV viral load ≥10,000 copies per mL of whole blood
7. Active infection with Cytomegalovirus (CMV) as defined by CMV viral load ≥10,000 copies per mL of whole blood
8. Diagnosis of liver disease or elevated hepatic enzymes, as defined by Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), or both > 1.5 x the upper limit of age-determined normal (ULN) or total bilirubin > ULN
9. Current or prior treatment that is known to cause a significant, ongoing change in the course of T1D or immunologic status
10. Current or prior (within last 30 days) use of drugs other than insulin to treat hyperglycemia (e.g. metformin, sulfonylureas, glinides, thiazolidinediones, exenatide, liraglutide, Dipeptidyl peptidase-4 Intravenous (DPP-IV) inhibitors, or amylin)
11. Current use of any medication known to significantly influence glucose tolerance (e.g., atypical antipsychotics, diphenylhydantoin, niacin)
12. Any of the following hematologic abnormalities, confirmed by repeat tests:

    1. White blood count <3,000/microL or >14,000/microL
    2. Lymphocyte count <500/microL
    3. Platelet count <150,000 /microL
    4. Hemoglobin <8.5 g/dL
    5. . Neutrophil count <2,000 cells/microL.
13. Females who are pregnant, lactating, or planning on pregnancy during the 2- year study period
14. History or diagnoses of other autoimmune diseases with the exception of stable thyroid or celiac disease
15. History of alcohol, drug or chemical abuse within 1 year prior to study eligibility screening evaluation
16. Any medical or psychological condition that in the opinion of the principal investigator would interfere with safe completion of the trial
17. Prior participation in a clinical trial that could increase risks associated with this clinical trial
18. Receipt of live vaccine (e.g. varicella, measles, mumps, rubella, cold-attenuated intranasal influenza vaccine, bacillus Calmette-Guérin, and small pox) in the 6 weeks before randomization
19. High lipid levels (fasting Low-density lipoprotein (LDL) cholesterol ≥160 mg/dL)
20. History of significant allergy (e.g. anaphylaxis) to milk or soy proteins.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Greenbaum, Study Chair — Benaroya Research Institute at Virginia Mason: Diabetes Research Program; Jane Buckner, M.D., Study Chair — Benaroya Research Institute at Virginia Mason: Diabetes Research Program
Locations (19):
- United States (17):
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Yale University School of Medicine: Diabetes Endocrinology Research Center, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami: Diabetes Research Institute, Miami, Florida
  - University of South Florida: Diabetes Center, Tampa, Florida
  - Indiana University Health - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Harvard University, Joslin Diabetes Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Columbia University, Naomi Berrie Diabetes Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Sanford Research, Sioux Falls, South Dakota
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Benaroya Research Institute, Seattle, Washington
- Australia (2):
  - The Children's Hospital at Westmead: Kids Research Institute, Westmead, New South Wales
  - Lady Cilento Children's Hospital: Department of Endocrinology, South Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- [Derived] Greenbaum CJ, Serti E, Lambert K, Weiner LJ, Kanaparthi S, Lord S, Gitelman SE, Wilson DM, Gaglia JL, Griffin KJ, Russell WE, Raskin P, Moran A, Willi SM, Tsalikian E, DiMeglio LA, Herold KC, Moore WV, Goland R, Harris M, Craig ME, Schatz DA, Baidal DA, Rodriguez H, Utzschneider KM, Nel HJ, Soppe CL, Boyle KD, Cerosaletti K, Keyes-Elstein L, Long SA, Thomas R, McNamara JG, Buckner JH, Sanda S; ITN058AI EXTEND Study Team. IL-6 receptor blockade does not slow beta cell loss in new-onset type 1 diabetes. JCI Insight. 2021 Nov 8;6(21):e150074. doi: 10.1172/jci.insight.150074. PMID 34747368
- [Derived] Hundhausen C, Roth A, Whalen E, Chen J, Schneider A, Long SA, Wei S, Rawlings R, Kinsman M, Evanko SP, Wight TN, Greenbaum CJ, Cerosaletti K, Buckner JH. Enhanced T cell responses to IL-6 in type 1 diabetes are associated with early clinical disease and increased IL-6 receptor expression. Sci Transl Med. 2016 Sep 14;8(356):356ra119. doi: 10.1126/scitranslmed.aad9943. PMID 27629486
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org/
- See also: EXTEND's study-specific ITN website — http://www.extendstudy.org/about-extend

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened from February 11, 2015 to Jun 21, 2018 at 17 sites in the US and two sites in Australia. March 12, 2015 was the actual date on which the first participant was enrolled in this clinical study.
Pre-assignment Details: Before initiating the study in the pediatric group (6-17 years old), adults (18-45 years old) were randomized 2:1 to tocilizumab or placebo, respectively. After at least 30 adults completed 12 weeks of treatment, the Data and Safety Monitoring Board (DSMB) and FDA reviewed the available data and allowed the enrollment of children 6-17 years old.
Groups:
- Tocilizumab (TCZ) in Pediatric Participants: Participants received intravenous (IV) infusions of either 8.0 mg/kg (body weight >=30 kg) or 10.0 mg/kg (body weight <30kg) tocilizumab every 4 weeks for 24 weeks. The dose was capped at 800 mg. Pediatric participants were 6 to 17 years old inclusive.
- Placebo in Pediatric Participants: Participants received IV placebo infusions of saline of equal volume and appearance to the treatment. Pediatric participants were 6 to 17 years old inclusive.
- Tocilizumab (TCZ) in Adult Participants: Participants received intravenous (IV) infusions of either 8.0 mg/kg (body weight >=30 kg) or 10.0 mg/kg (body weight <30kg) tocilizumab every 4 weeks for 24 weeks. The dose was capped at 800 mg. Adult participants were 18 to 45 years old inclusive.
- Placebo in Adult Participants: Participants received IV placebo infusions of saline of equal volume and appearance to the treatment. Adult participants were 18 to 45 years old inclusive.
Period: Overall Study
Arm/Group | Tocilizumab (TCZ) in Pediatric Participants | Placebo in Pediatric Participants | Tocilizumab (TCZ) in Adult Participants | Placebo in Adult Participants
Started | 54 | 27 | 35 (1 randomized adult was never treated) | 20
Completed | 51 | 23 | 31 | 19
Not Completed | 3 | 4 | 4 | 1
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 1
Not completed — COVID-19 Related | 1 | 1 | 0 | 0
Not completed — Participant ill and could not be infused | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants in each cohort were randomized 2:1 to tocilizumab or placebo, respectively.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tocilizumab (TCZ) in Pediatric Participants | Placebo in Pediatric Participants | Tocilizumab (TCZ) in Adult Participants | Placebo in Adult Participants | Total
Number analyzed (Participants) | 54 | 27 | 35 | 20 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.1 (2.9) | 11.1 (2.5) | 27.9 (7.4) | 29.2 (9.3) | 18.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 12 | 12 | 7 | 57
  Male | 28 | 15 | 23 | 13 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 3 | 1 | 9
  Not Hispanic or Latino | 53 | 21 | 32 | 19 | 125
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 1 | 2 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 0 | 3
  White | 47 | 20 | 32 | 19 | 118
  More than one race | 2 | 2 | 1 | 0 | 5
  Unknown or Not Reported | 2 | 2 | 0 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 24 | 35 | 20 | 131
  Australia | 2 | 3 | 0 | 0 | 5
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is a person's weight in kilograms divided by the square of height in meters. For more information regarding BMI, visit the Centers for Disease Control and Prevention (CDC) website, "How Do I Interpret Body Mass Index Information" at:
  https://www.cdc.gov/healthyweight/assessing/bmi/index.html
  kg/m^2 | 19.8 (3.8) | 19.1 (3.3) | 24.2 (3.9) | 25.4 (3.5) | 21.6 (4.4)
2-hour C-peptide Mean Area Under the Curve (mAUC) Result in Response to Standardized Mixed Meal Tol [Mean (Standard Deviation); unit: pmol/mL] — C-peptide is released by the pancreas into the bloodstream in equal amounts to insulin and reflects how much insulin pancreatic beta cells are making. The MMTT was performed in the morning and blood samples for C-peptide collected at baseline (pre-meal) and various minutes post-meal. C-peptide AUC was calculated using the trapezoidal rule over the 2-hour time period. Results of the stimulated 2-hour (e.g., 120 minutes) post-meal C-peptide AUC are provided. Larger numbers are preferable (better) in these AUC results: more insulin being produced reflects less severe disease.
  pmol/mL | 0.73 (0.44) | 0.66 (0.32) | 0.77 (0.24) | 0.97 (0.69) | 0.76 (0.43)
Hemoglobin A1C (HbA1c) Level [Mean (Standard Deviation); unit: percent (%)] — Glycosylated hemoglobin (HbA1c) is a measure of the average plasma concentration of blood sugar (glucose) over the previous three months and measures the level of optimal management of underlying disease. An HbA1c of 5.6% or less is considered normal. HbA1c of 6.5% or higher is typical for individuals with Type 1 Diabetes mellitus (T1DM). The closer HbA1c levels are to normal, the better controlled the disease is.
  percent (%) | 6.79 (1.03) | 6.86 (0.55) | 6.48 (1.08) | 6.28 (0.73) | 6.65 (0.94)
Average Insulin Use Per Kilogram Body Weight [Mean (Standard Deviation); unit: Units per Kilogram Body Weight per Day] — The need to use exogenous insulin is an indication that the body is not producing enough endogenous insulin. Higher amounts of insulin use indicate higher disease activity.
  Units per Kilogram Body Weight per Day | 0.39 (0.24) | 0.38 (0.19) | 0.28 (0.15) | 0.30 (0.21) | 0.35 (0.21)
Days from Type 1 Diabetes Mellitus (T1DM) Diagnosis to Randomization [Mean (Standard Deviation); unit: Days] — Inclusion criteria included being diagnosed with type 1 diabetes within 100 days of enrollment. Diagnosis was based on the American Diabetes Association T1DM criteria.
  Days | 85.9 (15.5) | 83.9 (16.7) | 82.5 (13.6) | 84.6 (12.4) | 84.4 (14.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 2-Hour C-peptide Mean Area Under the Curve (mAUC) in Pediatric Participants
Description: C-peptide is a substance released by the pancreas into the bloodstream in equal amounts to insulin and reflects how much insulin pancreatic beta cells are making. The standardized MMTT evaluates whether beta cells are producing endogenous insulin. The MMTT was performed in the morning and blood samples for C-peptide collected at baseline (pre-meal) and 15, 30, 60, 90, 120, 150, 180, 210, and 240 minutes post-meal. C-peptide mAUC was calculated using the trapezoidal rule over the 2-hour time period. Larger numbers are preferable (better) in these mAUC results: more insulin being produced reflects less severe disease. C-peptide levels in the serum (e.g., mAUC following a standardized MMTT) compared to control group at 1 year post treatment initiation for the evaluation of investigational products intended to preserve endogenous beta-cell function in T1DM trials is recognized by the Center for Drug Evaluation and Research (CDER) at the FDA as a valid efficacy endpoint.
Time Frame: Baseline (Pre-treatment) to Week 52
Population: The modified intent to treat population includes all randomized participants who received any dose of assigned study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Tocilizumab (TCZ) in Pediatric Participants | Placebo in Pediatric Participants
Number analyzed (Participants) | 54 | 27
pmol/mL | -0.337 [-0.39 to -0.28] | -0.391 [-0.47 to -0.31]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Week 52; Primary imputation method used for missing Week 52 mAUC; Test type: Superiority; p = 0.277, ANCOVA — P-value comes from an analysis of covariance with outcome variable of change in mAUC from screening and covariates of treatment, screening mAUC, and age

2. Secondary Outcome: Change From Baseline in 2-Hour C-peptide Mean Area Under the Curve (mAUC)
Description: as for outcome 1
Time Frame: Baseline (Pre-treatment) to Weeks 24, 52, and 104
Population: Modified intent to treat population includes all randomized participants who received any dose of assigned study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/mL
Groups:
- Tocilizumab (TCZ) in Pooled Participants: Participants received intravenous (IV) infusions of either 8.0 mg/kg (body weight >=30 kg) or 10.0 mg/kg (body weight <30kg) tocilizumab every 4 weeks for 24 weeks. The dose was capped at 800 mg. Pooled participants are the pediatric and adult participants who received TCZ combined.
- Placebo in Pooled Participants: Participants received IV placebo infusions of saline of equal volume and appearance to the treatment. Pooled participants are the pediatric and adult participants who received placebo combined.
Arm/Group | Tocilizumab (TCZ) in Pediatric Participants | Placebo in Pediatric Participants | Tocilizumab (TCZ) in Adult Participants | Placebo in Adult Participants | Tocilizumab (TCZ) in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 54 | 27 | 34 | 20 | 88 | 47
pmol/mL
  Week 24: number analyzed (Participants) | 54 | 26 | 33 | 20 | 87 | 46
  Week 24 | -0.200 [-0.26 to -0.14] | -0.164 [-0.25 to -0.08] | -0.072 [-0.17 to 0.03] | -0.097 [-0.23 to 0.03] | -0.152 [-0.20 to -0.10] | -0.134 [-0.21 to -0.06]
  Week 52: number analyzed (Participants) | 53 | 25 | 33 | 20 | 86 | 45
  Week 52 | -0.339 [-0.40 to -0.28] | -0.397 [-0.48 to -0.31] | -0.186 [-0.29 to -0.08] | -0.267 [-0.40 to -0.13] | -0.287 [-0.34 to -0.23] | -0.328 [-0.41 to -0.25]
  Week 104: number analyzed (Participants) | 49 | 22 | 29 | 19 | 78 | 41
  Week 104 | -0.495 [-0.55 to -0.44] | -0.556 [-0.64 to -0.47] | -0.384 [-0.49 to -0.28] | -0.388 [-0.52 to -0.25] | -0.461 [-0.52 to -0.40] | -0.463 [-0.54 to -0.38]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Week 24; Test type: Superiority; p = 0.499, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Week 52; Test type: Superiority; p = 0.267, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Week 104; Test type: Superiority; p = 0.226, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Week 24; Test type: Superiority; p = 0.758, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Week 52; Test type: Superiority; p = 0.341, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Week 104; Test type: Superiority; p = 0.969, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Week 24; Test type: Superiority; p = 0.689, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Week 52; Test type: Superiority; p = 0.400, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Week 104; Test type: Superiority; p = 0.969, ANCOVA — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: 2-Hour C-peptide Mean Area Under the Curve (mAUC), Mixed Model
Description: as for outcome 1
Time Frame: Baseline (Pre-treatment), Weeks 12, 24, 39, 52, 78, and 104
Population: The modified intent to treat population includes all randomized participants who received any dose of assigned study treatment. The model only included subjects with at least 1 post-screening assessment. One mITT subject did not have a post-screening MMTT and this subject is not included.
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Tocilizumab (TCZ) in Pediatric Participants | Placebo in Pediatric Participants | Tocilizumab (TCZ) in Adult Participants | Placebo in Adult Participants | Tocilizumab (TCZ) in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 54 | 26 | 34 | 20 | 88 | 46
pmol/mL
  Week 12 | 0.60 [0.51 to 0.69] | 0.55 [0.42 to 0.68] | 0.72 [0.56 to 0.89] | 0.88 [0.67 to 1.09] | 0.65 [0.57 to 0.74] | 0.69 [0.57 to 0.81]
  Week 24 | 0.55 [0.46 to 0.63] | 0.49 [0.37 to 0.61] | 0.68 [0.52 to 0.84] | 0.83 [0.62 to 1.04] | 0.60 [0.52 to 0.69] | 0.63 [0.52 to 0.75]
  Week 39 | 0.48 [0.40 to 0.56] | 0.42 [0.30 to 0.53] | 0.63 [0.47 to 0.79] | 0.77 [0.56 to 0.98] | 0.54 [0.46 to 0.62] | 0.56 [0.45 to 0.67]
  Week 52 | 0.42 [0.34 to 0.50] | 0.35 [0.24 to 0.46] | 0.59 [0.43 to 0.75] | 0.72 [0.51 to 0.93] | 0.49 [0.41 to 0.57] | 0.50 [0.39 to 0.61]
  Week 78 | 0.30 [0.23 to 0.37] | 0.23 [0.12 to 0.33] | 0.50 [0.33 to 0.66] | 0.61 [0.40 to 0.82] | 0.38 [0.30 to 0.46] | 0.38 [0.28 to 0.49]
  Week 104 | 0.18 [0.11 to 0.25] | 0.10 [0.00 to 0.21] | 0.41 [0.24 to 0.58] | 0.50 [0.28 to 0.72] | 0.27 [0.19 to 0.35] | 0.27 [0.16 to 0.38]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Screening to Week 104; Test type: Superiority; p = 0.679, Longitudinal mixed model — P-value is for group difference in time trends from a longitudinal mixed effects model. Response variable was 2-hour C-peptide mAUC and covariates were treatment, study week, age, treatment*study week, age*study week; Random within-subject effects for intercept and study week were included assuming an unstructured covariance matrix
Statistical Analysis 2: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Screening to Week 104; Test type: Superiority; p = 0.373, Longitudinal mixed model — [p-value comment as in outcome 3, analysis 1]; Random within-subject effects for intercept and study week were included assuming an unstructured covariance matrix
Statistical Analysis 3: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Screening to Week 104; Test type: Superiority; p = 0.395, Longitudinal mixed model — [p-value comment as in outcome 3, analysis 1]; Random within-subject effects for intercept and study week were included assuming an unstructured covariance matrix

4. Secondary Outcome: Change From Baseline in 4-Hour C-peptide Mean Area Under the Curve (mAUC)
Description: C-peptide is a substance released by the pancreas into the bloodstream in equal amounts to insulin and reflects how much insulin pancreatic beta cells are making. The standardized MMTT evaluates whether beta cells are producing endogenous insulin. The MMTT was performed in the morning and blood samples for C-peptide collected at baseline (pre-meal) and 15, 30, 60, 90, 120, 150, 180, 210, and 240 minutes post-meal. C-peptide mAUC was calculated using the trapezoidal rule over the 4-hour time period. Larger numbers are preferable (better) in these mAUC results: more insulin being produced reflects less severe disease. C-peptide levels in the serum (e.g., mAUC following a standardized MMTT) compared to control group at 1 year post treatment initiation for the evaluation of investigational products intended to preserve endogenous beta-cell function in T1DM trials is recognized by the Center for Drug Evaluation and Research (CDER) at the FDA as a valid efficacy endpoint.
Time Frame: Baseline (Pre-treatment) to Weeks 52 and 104
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Tocilizumab (TCZ) in Pediatric Participants | Placebo in Pediatric Participants | Tocilizumab (TCZ) in Adult Participants | Placebo in Adult Participants | Tocilizumab (TCZ) in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 54 | 27 | 34 | 20 | 88 | 47
pmol/mL
  Week 52: number analyzed (Participants) | 26 | 9 | 33 | 20 | 59 | 29
  Week 52 | -0.325 [-0.42 to -0.23] | -0.448 [-0.60 to -0.29] | -0.195 [-0.30 to -0.09] | -0.262 [-0.40 to -0.13] | -0.252 [-0.32 to -0.18] | -0.321 [-0.42 to -0.22]
  Week 104: number analyzed (Participants) | 24 | 7 | 29 | 19 | 53 | 26
  Week 104 | -0.521 [-0.62 to -0.42] | -0.635 [-0.82 to -0.45] | -0.382 [-0.49 to -0.27] | -0.390 [-0.53 to -0.25] | -0.449 [-0.53 to -0.37] | -0.448 [-0.56 to -0.33]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Week 52. Only participants >=12 years old had the 4-hour MMTT performed; Test type: Superiority; p = 0.176, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Week 104. Only participants >=12 years old had the 4-hour MMTT performed; Test type: Superiority; p = 0.285, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Week 52; Test type: Superiority; p = 0.435, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Week 104; Test type: Superiority; p = 0.931, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Week 52. Only participants >=12 years old had the 4-hour MMTT performed; Test type: Superiority; p = 0.280, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Week 104. Only participants >=12 years old had the 4-hour MMTT performed; Test type: Superiority; p = 0.985, ANCOVA — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline in Average Insulin Use in Units Per Kilogram Body Weight Per Day
Description: The need to use exogenous insulin is an indication that the body is not producing enough endogenous insulin. Higher amounts of insulin use indicate higher disease activity. Insulin use was collected each day for 5 days prior to the visit. Average insulin use per kg is the average insulin use over the 5 days prior to the visit divided by the participant's weight in kg.
Time Frame: Baseline (Pre-treatment) to Weeks 24, 52, and 104
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units per Kilogram Body Weight per Day
Arm/Group | Tocilizumab (TCZ) in Pediatric Participants | Placebo in Pediatric Participants | Tocilizumab (TCZ) in Adult Participants | Placebo in Adult Participants | Tocilizumab (TCZ) in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 54 | 27 | 34 | 20 | 88 | 47
Units per Kilogram Body Weight per Day
  Week 24: number analyzed (Participants) | 54 | 25 | 33 | 19 | 87 | 44
  Week 24 | 0.139 [0.09 to 0.19] | 0.126 [0.05 to 0.20] | 0.015 [-0.06 to 0.09] | 0.146 [0.05 to 0.24] | 0.090 [0.05 to 0.13] | 0.139 [0.08 to 0.20]
  Week 52: number analyzed (Participants) | 51 | 25 | 33 | 18 | 84 | 43
  Week 52 | 0.300 [0.24 to 0.36] | 0.326 [0.24 to 0.42] | 0.081 [0.01 to 0.15] | 0.112 [0.02 to 0.20] | 0.211 [0.16 to 0.26] | 0.243 [0.18 to 0.31]
  Week 104: number analyzed (Participants) | 50 | 23 | 30 | 17 | 80 | 40
  Week 104 | 0.403 [0.33 to 0.47] | 0.493 [0.39 to 0.59] | 0.116 [0.05 to 0.18] | 0.129 [0.05 to 0.21] | 0.288 [0.24 to 0.34] | 0.354 [0.28 to 0.43]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Week 24; Test type: Superiority; p = 0.762, ANCOVA — P-value comes from an analysis of covariance with outcome variable of change in average insulin use per kg from baseline and covariates of treatment, baseline average insulin use per kg, and age
Statistical Analysis 2: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Week 52; Test type: Superiority; p = 0.640, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Week 104; Test type: Superiority; p = 0.145, ANCOVA — P-value comes from an analysis of covariance with outcome variable of change in avg insulin use per kg from baseline and covariates of treatment, baseline average insulin use per kg, and age
Statistical Analysis 4: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Week 24; Test type: Superiority; p = 0.033, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Week 52; Test type: Superiority; p = 0.591, ANCOVA — P-value comes from an analysis of covariance with outcome variable of change in avg insulin use per kg from baseline and covariates of treatment, baseline avg insulin use per kg, and age
Statistical Analysis 6: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Week 104; Test type: Superiority; p = 0.810, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Week 24; Test type: Superiority; p = 0.178, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Week 52; Test type: Superiority; p = 0.430, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Week 104; Test type: Superiority; p = 0.149, ANCOVA — [p-value comment as in outcome 5, analysis 1]

6. Secondary Outcome: Change From Baseline in Average Insulin Use Per Kg, Mixed Model
Description: as for outcome 5
Time Frame: Baseline (Pre-treatment) to Weeks 12, 24, 39, 52, 78, and 104
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units per Kilogram Body Weight per Day
Arm/Group | Tocilizumab (TCZ) in Pediatric Participants | Placebo in Pediatric Participants | Tocilizumab (TCZ) in Adult Participants | Placebo in Adult Participants | Tocilizumab (TCZ) in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 54 | 27 | 34 | 20 | 88 | 47
Units per Kilogram Body Weight per Day
  Week 12 | 0.45 [0.40 to 0.51] | 0.45 [0.37 to 0.53] | 0.29 [0.22 to 0.35] | 0.37 [0.29 to 0.46] | 0.39 [0.35 to 0.43] | 0.42 [0.36 to 0.48]
  Week 24 | 0.50 [0.45 to 0.56] | 0.51 [0.44 to 0.59] | 0.31 [0.24 to 0.37] | 0.40 [0.31 to 0.48] | 0.43 [0.38 to 0.47] | 0.47 [0.41 to 0.53]
  Week 39 | 0.57 [0.51 to 0.62] | 0.59 [0.52 to 0.67] | 0.33 [0.26 to 0.40] | 0.43 [0.34 to 0.52] | 0.47 [0.43 to 0.52] | 0.53 [0.47 to 0.59]
  Week 52 | 0.62 [0.57 to 0.68] | 0.66 [0.58 to 0.74] | 0.35 [0.27 to 0.43] | 0.46 [0.36 to 0.56] | 0.51 [0.47 to 0.56] | 0.58 [0.52 to 0.64]
  Week 78 | 0.73 [0.67 to 0.79] | 0.80 [0.71 to 0.89] | 0.39 [0.30 to 0.49] | 0.51 [0.39 to 0.64] | 0.60 [0.54 to 0.65] | 0.68 [0.61 to 0.76]
  Week 104 | 0.84 [0.77 to 0.91] | 0.94 [0.83 to 1.04] | 0.43 [0.32 to 0.55] | 0.57 [0.42 to 0.72] | 0.68 [0.62 to 0.74] | 0.79 [0.70 to 0.87]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Screening to Week 104; Test type: Superiority; p = 0.103, Longitudinal mixed model — P-value is for group difference in time trends from a longitudinal mixed effects model. Response variable was average insulin use per kg and covariates were treatment, study week, age, treatment*study week, age*study week; Random within-subject effects for intercept and study week were included assuming an unstructured covariance matrix
Statistical Analysis 2: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Screening to Week 104; Test type: Superiority; p = 0.452, Longitudinal mixed model — [p-value comment as in outcome 6, analysis 1]; Random within-subject effects for intercept and study week were included assuming an unstructured covariance matrix
Statistical Analysis 3: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Screening to Week 104; Test type: Superiority; p = 0.091, Longitudinal mixed model — [p-value comment as in outcome 6, analysis 1]; Random within-subject effects for intercept and study week were included assuming an unstructured covariance matrix

7. Secondary Outcome: Change From Baseline in Hemoglobin A1c
Description: Glycosylated hemoglobin (HbA1c) is a measure of the average plasma concentration of blood sugar (glucose) over the previous three months and measures the level of optimal management of underlying disease. An HbA1c of 5.6% or less is considered normal. HbA1c of 6.5% or higher is typical for individuals with Type 1 Diabetes mellitus (T1DM). The closer HbA1c levels are to normal, the better controlled the disease is.
Time Frame: Baseline (Pre-treatment) to Weeks 24, 52, and 104
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent (%)
Arm/Group | Tocilizumab (TCZ) in Pediatric Participants | Placebo in Pediatric Participants | Tocilizumab (TCZ) in Adult Participants | Placebo in Adult Participants | Tocilizumab (TCZ) in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 54 | 27 | 34 | 20 | 88 | 47
percent (%)
  Week 24: number analyzed (Participants) | 54 | 26 | 33 | 20 | 87 | 46
  Week 24 | 0.065 [-0.17 to 0.30] | 0.368 [0.02 to 0.71] | -0.509 [-0.80 to -0.21] | -0.136 [-0.51 to 0.24] | -0.163 [-0.34 to 0.02] | 0.169 [-0.08 to 0.42]
  Week 52: number analyzed (Participants) | 53 | 25 | 32 | 20 | 85 | 45
  Week 52 | 0.650 [0.24 to 1.06] | 1.134 [0.53 to 1.74] | 0.152 [-0.21 to 0.51] | 0.262 [-0.19 to 0.72] | 0.459 [0.16 to 0.76] | 0.753 [0.34 to 1.17]
  Week 104: number analyzed (Participants) | 49 | 22 | 31 | 19 | 80 | 41
  Week 104 | 0.734 [0.33 to 1.14] | 1.042 [0.44 to 1.64] | 0.253 [-0.21 to 0.71] | 0.583 [0.00 to 1.17] | 0.556 [0.25 to 0.86] | 0.812 [0.38 to 1.24]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Week 24; Test type: Superiority; p = 0.154, ANCOVA — P-value comes from an analysis of covariance with outcome variable of change in HbA1c from baseline and covariates of treatment, baseline HbA1c, and age
Statistical Analysis 2: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Week 52; Test type: Superiority; p = 0.193, ANCOVA — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Week 104; Test type: Superiority; p = 0.397, ANCOVA — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Week 24; Test type: Superiority; p = 0.125, ANCOVA — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Week 52; Test type: Superiority; p = 0.705, ANCOVA — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 6: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Week 104; Test type: Superiority; p = 0.378, ANCOVA — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 7: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Week 24; Test type: Superiority; p = 0.035, ANCOVA — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 8: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Week 52; Test type: Superiority; p = 0.262, ANCOVA — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 9: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Week 104; Test type: Superiority; p = 0.338, ANCOVA — [p-value comment as in outcome 7, analysis 1]

8. Secondary Outcome: Change From Baseline in Hemoglobin A1C (HbA1c) Level in Participants, Mixed Model
Description: as for outcome 7
Time Frame: Baseline (Pre-treatment) to Weeks 12, 24, 39, 52, 78, and 104
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent (%)
Arm/Group | Tocilizumab (TCZ) in Pediatric Participants | Placebo in Pediatric Participants | Tocilizumab (TCZ) in Adult Participants | Placebo in Adult Participants | Tocilizumab (TCZ) in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 54 | 27 | 34 | 20 | 88 | 47
percent (%)
  Week 12 | 6.74 [6.50 to 6.97] | 6.99 [6.65 to 7.32] | 5.88 [5.59 to 6.18] | 6.04 [5.65 to 6.43] | 6.40 [6.21 to 6.58] | 6.60 [6.35 to 6.86]
  Week 24 | 6.87 [6.65 to 7.10] | 7.20 [6.88 to 7.52] | 6.02 [5.71 to 6.34] | 6.19 [5.78 to 6.60] | 6.54 [6.35 to 6.72] | 6.79 [6.54 to 7.04]
  Week 39 | 7.05 [6.80 to 7.29] | 7.46 [7.11 to 7.82] | 6.19 [5.85 to 6.54] | 6.38 [5.93 to 6.83] | 6.71 [6.51 to 6.91] | 7.02 [6.75 to 7.30]
  Week 52 | 7.20 [6.91 to 7.48] | 7.69 [7.28 to 8.11] | 6.34 [5.96 to 6.73] | 6.54 [6.04 to 7.03] | 6.86 [6.63 to 7.09] | 7.23 [6.91 to 7.54]
  Week 78 | 7.50 [7.10 to 7.90] | 8.16 [7.57 to 8.74] | 6.64 [6.17 to 7.11] | 6.86 [6.26 to 7.47] | 7.16 [6.85 to 7.46] | 7.63 [7.21 to 8.05]
  Week 104 | 7.80 [7.26 to 8.34] | 8.62 [7.83 to 9.40] | 6.94 [6.37 to 7.51] | 7.19 [6.45 to 7.92] | 7.45 [7.06 to 7.85] | 8.04 [7.49 to 8.59]
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Screening to Week 104; Test type: Superiority; p = 0.493, Longitudinal mixed model — P-value is for group difference in time trends from a longitudinal mixed effects model. Response variable was HbA1c and covariates were treatment, study week, spline week (at week 4), age, treatment*spline week, treatment*study week, age*study week; Random within-subject effects for intercept, study week, and spline week were included assuming an unstructured covariance matrix
Statistical Analysis 2: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Screening to Week 104; Test type: Superiority; p = 0.659, Longitudinal mixed model — [p-value comment as in outcome 8, analysis 1]; [statistical method as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Screening to Week 104; Test type: Superiority; p = 0.407, Longitudinal mixed model — [p-value comment as in outcome 8, analysis 1]; [statistical method as in outcome 8, analysis 1]

9. Secondary Outcome: Number of Participants Who Experienced at Least One Major Hypoglycemic Event After Treatment Initiation
Description: Major hypoglycemic adverse events are defined as: Blood glucose concentration < 40 mg/dL (Grades 3-5, NCI-CTCAE version 4.03*), or hypoglycemic events involving seizure or loss of consciousness (coma) or requiring assistance from another individual in order to recover.
  *NCI-CTCAE: National Cancer Institute Common Terminology Criteria for Adverse Events
Time Frame: Day 0 (Treatment Initiation) to Weeks 52 and 104
Population: The safety population includes all participants who received any degree of study treatment. Safety analyses are based on actual treatment the participants receive.
Measure: Number; unit: Participants
Arm/Group | Tocilizumab (TCZ) in Pediatric Participants | Placebo in Pediatric Participants | Tocilizumab (TCZ) in Adult Participants | Placebo in Adult Participants | Tocilizumab (TCZ) in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 54 | 27 | 34 | 20 | 88 | 47
Participants
  Day 0 to Week 52 | 19 | 11 | 10 | 3 | 29 | 14
  Day 0 to Week 104 | 28 | 14 | 15 | 8 | 43 | 22
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Baseline to Week 52; Test type: Superiority; p = 0.634, Fisher Exact — P-value is from comparing the number of participants with a hypoglycemic event between the two treatment groups using Fisher's exact test
Statistical Analysis 2: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Baseline to Week 104/End of Study; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Baseline to Week 52; Test type: Superiority; p = 0.329, Fisher Exact — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Baseline to Week 104/End of Study; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Baseline to Week 52; Test type: Superiority; p = 0.847, Fisher Exact — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Baseline to Week 104/End of Study; Test type: Superiority; p = 0.858, Fisher Exact — [p-value comment as in outcome 9, analysis 1]

10. Secondary Outcome: Number of Participants Who Experienced Infusion-Related Adverse Events
Description: An infusion/dose reaction is defined as an adverse event occurring during and within 24 hours after the infusion or subcutaneous injection of tocilizumab. This may include hypersensitivity reactions or anaphylactic reactions.
Time Frame: Day 0 (Treatment Initiation) to Week 52
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Tocilizumab (TCZ) in Pediatric Participants | Placebo in Pediatric Participants | Tocilizumab (TCZ) in Adult Participants | Placebo in Adult Participants | Tocilizumab (TCZ) in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 54 | 27 | 34 | 20 | 88 | 47
Participants | 4 | 0 | 5 | 0 | 9 | 0
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Treatment start to Week 52; Test type: Superiority; p = 0.296, Fisher Exact — P-value is from comparing the number of participants with the AEs of interest between the two treatment groups using Fisher's exact test
Statistical Analysis 2: Comparison: Tocilizumab (TCZ) in Adult Participants vs Placebo in Adult Participants; Treatment start to Week 52; Test type: Superiority; p = 0.145, Fisher Exact — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Treatment start to Week 52; Test type: Superiority; p = 0.027, Fisher Exact — [p-value comment as in outcome 10, analysis 1]

11. Secondary Outcome: Number of Participants Who Experienced Hypersensitivity Adverse Events
Description: Signs of a possible hypersensitivity reaction to the study drug include but are not limited to:
  * Fever, chills, pruritus, urticaria, angioedema, and skin rash
  * Cardiopulmonary reactions, including chest pain, dyspnea, hypotension or hypertension
Time Frame: Day 0 (Treatment Initiation) to Week 52
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Tocilizumab (TCZ) in Pediatric Participants | Placebo in Pediatric Participants | Tocilizumab (TCZ) in Adult Participants | Placebo in Adult Participants | Tocilizumab (TCZ) in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 54 | 27 | 34 | 20 | 88 | 47
Participants | 3 | 0 | 0 | 0 | 3 | 0
Statistical Analysis 1: Comparison: Tocilizumab (TCZ) in Pediatric Participants vs Placebo in Pediatric Participants; Treatment start to Week 52; Test type: Superiority; p = 0.547, Fisher Exact — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Tocilizumab (TCZ) in Pooled Participants vs Placebo in Pooled Participants; Treatment start to Week 52; Test type: Superiority; p = 0.551, Fisher Exact — [p-value comment as in outcome 10, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 104 weeks.
Arm/Group | Tocilizumab (TCZ) in Pediatric Participants | Placebo in Pediatric Participants | Tocilizumab (TCZ) in Adult Participants | Placebo in Adult Participants | Tocilizumab (TCZ) in Pooled Participants | Placebo in Pooled Participants
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/27 | 0/34 | 0/20 | 0/88 | 0/27
Serious Adverse Events (participants affected / at risk) | 3/54 | 3/27 | 2/34 | 2/20 | 5/88 | 5/47
Other Adverse Events (participants affected / at risk) | 52/54 | 26/27 | 31/34 | 19/20 | 83/88 | 45/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (TCZ) in Pediatric Participants (N=54) | Placebo in Pediatric Participants (N=27) | Tocilizumab (TCZ) in Adult Participants (N=34) | Placebo in Adult Participants (N=20) | Tocilizumab (TCZ) in Pooled Participants (N=88) | Placebo in Pooled Participants (N=47)
Vaccination site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thoracic outlet syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (TCZ) in Pediatric Participants (N=54) | Placebo in Pediatric Participants (N=27) | Tocilizumab (TCZ) in Adult Participants (N=34) | Placebo in Adult Participants (N=20) | Tocilizumab (TCZ) in Pooled Participants (N=88) | Placebo in Pooled Participants (N=47)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 1 (1)
Basedow's disease (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 3 (4) | 0 (0) | 1 (1) | 2 (3) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 5 (7) | 3 (4) | 2 (2) | 0 (0) | 7 (9) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 4 (4) | 4 (4)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 1 (1) | 4 (4) | 3 (3) | 8 (9) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1) | 2 (3) | 4 (4) | 6 (7)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (20) | 4 (11) | 5 (8) | 2 (2) | 18 (28) | 6 (13)
Vomiting (Gastrointestinal disorders) | 10 (16) | 6 (7) | 4 (4) | 1 (1) | 14 (20) | 7 (8)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Influenza like illness (General disorders) | 1 (1) | 3 (5) | 2 (3) | 2 (2) | 3 (4) | 5 (7)
Pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 7 (9) | 4 (5) | 1 (1) | 0 (0) | 8 (10) | 4 (5)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 6 (7) | 2 (3) | 0 (0) | 2 (2) | 6 (7) | 4 (5)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
Ear infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 9 (9) | 3 (3) | 6 (6) | 2 (6) | 15 (15) | 5 (9)
Gastroenteritis viral (Infections and infestations) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 1 (1)
Influenza (Infections and infestations) | 8 (8) | 5 (5) | 1 (1) | 2 (2) | 9 (9) | 7 (7)
Nasopharyngitis (Infections and infestations) | 7 (10) | 4 (6) | 5 (10) | 2 (2) | 12 (20) | 6 (8)
Oral herpes (Infections and infestations) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (4) | 1 (1)
Otitis externa (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Otitis media (Infections and infestations) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 3 (3)
Pharyngitis (Infections and infestations) | 5 (6) | 3 (4) | 4 (4) | 0 (0) | 9 (10) | 3 (4)
Pharyngitis streptococcal (Infections and infestations) | 6 (6) | 0 (0) | 0 (0) | 1 (2) | 6 (6) | 1 (2)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Sinusitis (Infections and infestations) | 5 (11) | 1 (3) | 4 (4) | 0 (0) | 9 (15) | 1 (3)
Skin infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 26 (82) | 13 (35) | 15 (42) | 12 (30) | 41 (124) | 25 (65)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 5 (6) | 3 (3) | 5 (6) | 4 (4)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 3 (6) | 0 (0) | 1 (1) | 0 (0) | 4 (7) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Body mass index increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 3 (5) | 0 (0) | 5 (7) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 28 (85) | 14 (47) | 15 (42) | 7 (11) | 43 (127) | 21 (58)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 4 (4) | 4 (8) | 7 (8) | 4 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 5 (5) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (2) | 3 (3) | 2 (5) | 7 (7) | 3 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 4 (5) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 2 (4) | 4 (4) | 1 (1) | 6 (6) | 3 (5)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 14 (24) | 6 (17) | 5 (8) | 6 (7) | 19 (32) | 12 (24)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 3 (4) | 2 (2) | 1 (1) | 3 (3) | 4 (5)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 5 (5) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (9) | 2 (4) | 2 (2) | 11 (13) | 9 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2) | 4 (4) | 3 (3) | 8 (10) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (17) | 4 (5) | 5 (6) | 1 (1) | 14 (23) | 5 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 4 (4)
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (8) | 0 (0) | 2 (8) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (2) | 0 (0) | 0 (0) | 3 (5) | 1 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 5 (5) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 2 (2) | 1 (1) | 4 (4) | 5 (6)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (4) | 5 (5) | 2 (2) | 12 (13) | 5 (6)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Family stress (Social circumstances) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT02293837/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT02293837/SAP_001.pdf